CLINICAL TRIAL: NCT06988813
Title: Bidirectional Cohort Study of Nanfang Spondyloarthritis
Acronym: BCNS
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-228
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Spondyloarthritis (SpA); Ankylosing Spondylitis (AS)
Keywords: Bidirectional Cohort
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: Patients between May 2024 and April 2025 were required to sign an up-to-date Ethics Committee-approved Informed Consent Form (ICF) prior to data collection, and all clinical data were collected at once. Patients with visits from April 2010 to April 2024 (and who will not return to the hospital at a later date) will be exempted from informed consent for this study, as the information involved in the visit will come from the medical record of the clinical visit, the risk to the subject is no more than minimal, the exemption from informed consent will not adversely affect the patient's rights or health and the study will not be able to proceed if informed consent is obtained, and subjects' privacy and personally identifiable information will be protected. Subjects' privacy and personally identifiable information will be protected.
- Prospective cohort: Patients will be required to sign an up-to-date Ethics Committee-approved Informed Consent Form (ICF) prior to data collection. After obtaining informed consent from patients, information on routine clinical visits will be collected, and the number and timing of study visits will follow the time points for routine clinical patient review. The time points for routine clinical review will be: every 3 months for 1 year and every 6 months for 3 years after treatment, for a total of 4 years.

SUMMARY:
Spondyloarthritis（SpA） patients attending Nanfang Hospital of Southern Medical University will generate a large number of clinical condition scales, laboratory indicators, imaging data such as X-rays or MRIs in the course of multiple standardized follow-up visits, as well as medical specimens from some of the patients who undergo surgical treatments. The Department of Orthopaedic Surgery of Nanfang Hospital is looking forward to the future and proposes to establish a specialized cohort named "Nanfang SpA Bidirectional Specialized Disease Cohort" by simply recording the clinical and imaging data of the above patients who have attended the clinic, been treated routinely, and have been followed up in the department without any interventional research measures. The cohort is proposed to: (1) archive the disease characteristics, biochemical index data, and disease assessment scales of all SpA patients attending the Southern Hospital; (2) record the X-ray and magnetic resonance imaging data of the patients to establish the "Southern SpA Imaging Dataset". This provides strong support for subsequent SpA research projects and lays the foundation for subsequent large-scale transect studies and retrospective studies.

DETAILED DESCRIPTION:
In this study, on the basis of not imposing randomized or interventional treatments and not generating additional examination tests on patients, the chronic disease data formed by multiple visits of SpA patients using conventional treatment regimens were used to form a bi-directional, disease-specific cohort by means of data entry alone, consisting of: one SpA condition information dataset, one SpA imaging dataset.

SpA condition information dataset: enter the disease duration, symptom characteristics, family history, comorbidities, previous medication use and efficacy of all outpatient diagnosed SpA patients; for each natural visit time point, establish BASDAI and ASDASCRP scores to assess the disease activity, assess the patient's physical functioning by BASFI scale, and EQ-5D and SF-36 scales to assess the quality of life; Recorded labs for each visit such as CRP, ESR and anti-streptococcal hemolysin O (ASO), anti-streptococcal DNAase B (ADNS). The subject group will not direct patients to lab tests that are not prescribed by the attending physician.

SpA imaging dataset: all imaging data of patients diagnosed with SpA and naturally attending our clinic were recorded, including: MRI of sacroiliac joints, MRI of hips, MRI of cervical/lumbar/thoracic spine, and orthopantomogram of pelvis, CT of sacroiliac joints, or vascular ultrasound of sacroiliac joints and lower limbs, and the imaging data were archived after preliminary SPARCC and SPARCC SSS scores were made. The subject group would not direct patients to examinations that were not prescribed by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* 1.Attended Nanfang Hospital, Southern Medical University, 2010-2030 2.Prospective cohort study component: subjects voluntarily participate with informed consent and sign an informed consent form 3.Retrospective cohort study: (i) patients who visited the hospital from April 2010 to April 2024 (and who will not return to the hospital at a later date) were exempted from informed consent; (ii) patients who visited the hospital from May 2024 to April 2025 were required to sign an informed consent 4.10 years old ≤ age ≤ 59 years old 5.Patients with a standardized diagnosis of spondyloarthritis by the following guidelines or diagnostic criteria, i.e., meeting one of the following diagnostic criteria: (1) 2009 ASAS classification criteria for axial spondyloarthritis; (2) 2011 ASAS classification criteria for peripheral spondyloarthritis

Exclusion Criteria:

* 1. Women who are pregnant, preparing for pregnancy or breastfeeding 2.Moderate to Severe Heart Failure (New York Heart Association Class 3-4) 3.Active peptic ulcers/bleeding 4.Judged by the investigator to be unsuitable for participation in this study

Ages: 10 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Spondyloarthritis (SpA) is a group of diseases characterized by inflammation of the sacro-skeletal joints and the tendon attachment points of the spine and peripheral joints, etc. The course of SpA is characterized by gradual progression, and it is divided into three main stages, from mild to severe, namely, undifferentiated SpA (uSpA), sacroiliac arthritis, and AS. The uSpA stage is characterized by a gradual progression.In the uSpA stage, the only manifestations are fat metaplasia or inflammation of the attachment points of the sacroiliac joints, while in the sacroiliac arthritis stage, subchondral intramedullary edema of the sacroiliac joints develops, and in the AS stage, sacroiliac erosion and fusion of the joints occur.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-05-17 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
SpA dateset | From enrollment to the end of the follow-up at the 48th week
  Collect a proprietary profile of clinical characteristics, laboratory and scale data, and imaging images from the Southern SpA Bi-directional Cohort for investigators to understand the natural history of the disease and to identify risk and prognostic factors for SpA.

SECONDARY OUTCOMES:
Disease activity score | From the start of enrollment, the follow-up time point was once every 3 months within the first year, and then once every 6 months within the subsequent 3 years
  These include: Patient's Global Assessment, Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score, C-reactive protein-based Ankylosing Spondylitis Disease Activity Score (ASDASCRP score), Bath Ankylosing Spondylitis Measurement Index (BASMI) score, Maastricht Ankylosing Spondylitis Attachment Spondylitis (MASES) score, Swollen Joint Count (Swollen Joint Count, 44 joint counts), Tender Joint Count (Tender Joint Count) (ASDASCRP score), Maastricht Ankylosing Spondylitis Attachment Spondylitis (MASES) score, Swollen Joint Count (Swollen Joint Count, 44 joints counted), Tender Joint Count (Tender Joint Count, 46 joints counted).
Quality of life score | From the start of enrollment, the follow-up time point was once every 3 months within the first year, and then once every 6 months within the subsequent 3 years
  These include: Bath Ankylosing Spondylitis Functional Index (BASFI) Score, Quality of Survival Measurement for Ankylosing Spondylitis Patients (SQOL-AS), Short Form Health Survey (SF-36), BAS-G Score, Health Questionnaire for Spondyloarthritis (HAQ-S), Questionnaire of Productivity and Activity Impairment for Specific Health Problems (WPAI-SHP).
Imaging Evaluation | From the start of enrollment, the follow-up time point was once every 3 months within the first year, and then once every 6 months within the subsequent 3 years
  Assessment of the severity of the condition on imaging (e.g., X-ray or MRI), such as: sacroiliac pathologic changes using the Spondyloarthritis Research Consortium of Canada Score(SPARCC), and spinal lesions using the Modified Stoke Ankylosing Spondylitis Spine Score(mSASSS).
Adverse events | From the start of enrollment, the follow-up time point was once every 3 months within the first year, and then once every 6 months within the subsequent 3 years
  Record the type, frequency, and severity of all treatment-related adverse events, and use CTCAE criteria to categorize them for a comprehensive assessment of the safety of the consultation process.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hostipal,Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided